CLINICAL TRIAL: NCT07318883
Title: A Randomized, Double-Blind, Multicenter, Phase II/III Clinical Study to Evaluate HLX07 (Recombinant Anti-EGFR Humanized Monoclonal Antibody Injection) in Combination With Serplulimab and Chemotherapy Versus Placebo in Combination With Serplulimab or Pembrolizumab and Chemotherapy as First-Line Treatment in Patients With Advanced Squamous Non-Small Cell Lung Cancer (sqNSCLC)
Brief Title: A Phase II/III Clinical Study to Evaluate HLX07 in Combination With Serplulimab and Chemotherapy Versus Placebo in Combination With Serplulimab or Pembrolizumab and Chemotherapy as First-Line Treatment in Advanced Squamous Non-Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX07-sqNSCLC301
Record Dates: First submitted 2026-01-04; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Squamous NSCLC
MeSH Terms: interventions — HLX07; pembrolizumab; Carboplatin; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part I (phase 2)-Group A (Experimental): HLX07 + serplulimab + carboplatin + paclitaxel or nab-paclitaxel, once every 3 weeks for a total of 4 cycles, followed by maintenance therapy with HLX07 in combination with serplulimab, with serplulimab administered for up to 2 years.
  Interventions: Drug: HLX07; Drug: Serplulimab; Drug: Carboplatin; Drug: Paclitaxel or Nab-Paclitaxel
- Part I (phase 2)-Group B (Active Comparator): Placebo + serplulimab + carboplatin + paclitaxel or nab-paclitaxel, once every 3 weeks for a total of 4 cycles, followed by maintenance therapy with placebo in combination with serplulimab, with serplulimab administered for up to 2 years.
  Interventions: Drug: HLX07 placebo; Drug: Serplulimab; Drug: Carboplatin; Drug: Paclitaxel or Nab-Paclitaxel
- Part II (phase 3)-Group A (Experimental): HLX07 + serplulimab + carboplatin + paclitaxel or nab-paclitaxel, once every 3 weeks for a total of 4 cycles, followed by maintenance therapy with HLX07 in combination with serplulimab, with serplulimab administered for up to 2 years.
  Interventions: Drug: HLX07; Drug: Serplulimab; Drug: Carboplatin; Drug: Paclitaxel or Nab-Paclitaxel
- Part II (phase 3)-Group B (Active Comparator): Placebo + pembrolizumab + carboplatin + paclitaxel or nab-paclitaxel, once every 3 weeks for a total of 4 cycles, followed by maintenance therapy with placebo in combination with pembrolizumab, with pembrolizumab administered for up to 2 years.
  Interventions: Drug: HLX07 placebo; Drug: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel or Nab-Paclitaxel

INTERVENTIONS:
Drug: HLX07 — Intravenous infusion (IV), once every 3 weeks (Day 1 of each cycle [D1]).
  Arms: Part I (phase 2)-Group A; Part II (phase 3)-Group A
Drug: HLX07 placebo — Intravenous infusion (IV), once every 3 weeks (Day 1 of each cycle [D1]).
  Arms: Part I (phase 2)-Group B; Part II (phase 3)-Group B
Drug: Serplulimab — IV, once every 3 weeks (D1).
  Other Names: HLX10
  Arms: Part I (phase 2)-Group A; Part I (phase 2)-Group B; Part II (phase 3)-Group A
Drug: Pembrolizumab — IV, once every 3 weeks (D1).
  Other Names: Keytruda
  Arms: Part II (phase 3)-Group B
Drug: Carboplatin — IV, once every 3 weeks (D1).
Drug: Paclitaxel or Nab-Paclitaxel — Paclitaxel: IV, once every 3 weeks (D1). Nab-paclitaxel: IV, once every 3 weeks (D1, 8, 15).

SUMMARY:
The study consists of two parts:

Part I is a randomized, double-blind, multicenter, parallel-controlled phase II clinical study to evaluate the efficacy and safety of HLX07 in combination with serplulimab and chemotherapy versus placebo in combination with serplulimab and chemotherapy as first-line treatment in patients with sqNSCLC.

Part II is a randomized, double-blind, multicenter, parallel-controlled phase III clinical study to evaluate the efficacy and safety of HLX07 in combination with serplulimab and chemotherapy versus placebo in combination with pembrolizumab and chemotherapy as first-line treatment in patients with sqNSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. The patients voluntarily participate in this clinical study, fully understand and have been informed about the study, have signed the informed consent form (ICF), and are willing to follow and able to complete all study procedures.
2. Male or female, aged 18 years or older at the time of signing the ICF.
3. Histologically confirmed with stage IIIB/IIIC or IV (AJCC 8th edition) squamous NSCLC ineligible for surgery or radical radiotherapy.
4. Patients must provide sufficient tumor tissues that meet the quality requirements for the determination of EGFR and PD-L1 expression levels.

   Note: Formalin-fixed tumor samples (paraffin blocks or unstained sections, meeting the quality control criteria for testing) collected from lesions that have not received radiotherapy at or after the diagnosis of locally advanced/recurrent or distant metastatic squamous non-small cell lung cancer (sqNSCLC) (from the most recent surgery or biopsy, preferably within half a year prior to randomization) should be provided. Relevant pathology reports must also be provided for the above specimens. For detailed requirements for tissue samples, see the Laboratory Operation Manual.
5. Absence of prior systemic treatment for locally advanced/recurrent or distant metastatic sqNSCLC. Patients who have received prior adjuvant or neoadjuvant therapy are allowed to be enrolled if the adjuvant/neoadjuvant therapy has been completed at least 6 months before the diagnosis of locally advanced/recurrent or distant metastatic sqNSCLC.
6. Prior non-systemic anti-tumor therapy or Chinese herbal anti-tumor therapy must have ended for ≥ 2 weeks before randomization, and treatment-related AEs have resolved to Grade ≤ 1 according to Common Terminology Criteria for Adverse Events (CTCAE) 6.0 (except for Grade 2 alopecia).
7. At least one measurable target lesion assessed by BICR as per RECIST v1.1 within 4 weeks before randomization.

   Note: Measurable target lesions cannot be selected from prior radiotherapy sites. A lesion at the prior radiotherapy site may be selected as the target lesion if it is the only available lesion, and should provide the imaging data of the lesion before and after an unequivocal progression after the radiotherapy.
8. An ECOG performance status score of 0 or 1 within 7 days prior to randomization.
9. Life expectancy ≥ 12 weeks.
10. Hepatitis B surface antigen (HBsAg) (-) and hepatitis B core antibody (HBcAb) (-); if HBsAg (+) or HBcAb (+), hepatitis B virus deoxyribonucleic acid (HBV-DNA) must be < 2,500 copies/mL or 500 IU/mL or within the normal range of this site.
11. HCV antibody (-); if HCV antibody (+), HCV-RNA testing must be negative before enrollment. Participants co-infected with hepatitis B and C will be excluded (tested positive for HBsAg or HBcAb and positive for HCV antibody).
12. Adequate major organ functions as defined by the following criteria
13. Female patients must meet one of the following conditions:

    * Post-menopausal (defined as amenorrhea for at least 1 year with no documented cause other than menopause), or
    * Surgically sterilized (removal of the ovaries and/or uterus), or
    * Fertile, but must:

      * be tested negative for serum pregnancy test within 7 days prior to randomization, and
      * agree to use contraception with an annual failure rate of < 1% or to remain abstinent (avoid heterosexual intercourse) from signing the informed consent form to at least 6 months after the last dose of study drugs (contraception with an annual failure rate of < 1% includes bilateral tubal ligation, male sterilization, correct use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper-containing intrauterine devices), and not donate eggs during this period, and
      * not breastfeed.
14. Male patients must: agree to remain abstinent (avoid heterosexual intercourse) or take contraception measures as follows: male patients with a pregnant partner or a partner with childbearing potential must remain abstinent or take contraception measures for contraception during the treatment period with the study drugs and for at least 6 months after the last dose to prevent the drug exposure to the embryo. Periodic abstinence (e.g., contraception based on calendar day, ovulatory phase, basal body temperature, or postovulatory phase) and external ejaculation are ineligible methods of contraception. Sperm donation is prohibited during this period.
15. Patients who have previously received denosumab and are eligible for and agree to switch to bisphosphonates for bone metastases.

Exclusion Criteria:

1. Histologically confirmed non-sqNSCLC. Mixed tumors will be classified by the predominant cell type. Patients with small cell component or neuroendocrine carcinoma component are not eligible. For the non-small cell histology, patients with squamous component that is predominant (e.g., adenosquamous) are eligible.
2. Known EGFR-sensitizing mutation, ALK/ROS1 gene rearrangement, or other actionable driver oncogenes for which there are locally approved targeted first-line therapies.

   Note: If the EGFR, ALK, ROS1 and other actionable driver oncogenes statuses are unknown, testing is not mandatory, unless there are high-risk factors (such as non-smoking female patients), under which circumstances testing of EGFR and other mutations may be considered.
3. Other malignancies within 5 years or active. Patients with localized tumors that have been cured, such as basal cell carcinoma, squamous-cell skin cancer, superficial bladder carcinoma, prostate carcinoma in situ, cervical carcinoma in situ, and breast cancer in situ, are eligible.
4. Scheduled or previous organ or bone marrow transplantation.
5. Uncontrollable pleural effusion, pericardial effusion, or ascites.
6. Active central nervous system (CNS) metastases and/or carcinomatous meningitis known or diagnosed at screening. However, the following patients may be enrolled:

   * Patients with asymptomatic brain metastases (i.e., no progressive central nervous system symptoms caused by brain metastases, no requirement for glucocorticoid therapy, and lesion size ≤ 1.5 cm) may be enrolled, but are required to receive regular brain imaging as a site of lesion.
   * Patients with treated brain metastases that have been stable for at least 1 month, with no evidence of new or enlarging brain metastases, and with glucocorticoid discontinued ≥ 3 days prior to randomization.

   Stable brain metastases should be confirmed before randomization.
7. Spinal cord compression that has not been cured with radical surgery and/or radiotherapy.
8. Clinically significant hemoptysis complicated with superior vena cava syndrome.
9. Myocardial infarction and poorly controlled arrhythmia (including QTc intervals ≥ 450 ms for males and ≥ 470 ms for females) (QTc intervals are calculated by Fridericia's formula) within 6 months prior to randomization;
10. NYHA Class III-IV cardiac insufficiency or left ventricular ejection fraction (LVEF) < 50% by echocardiography.
11. Inadequately controlled hypertension (defined as systolic blood pressure ≥ 150 mmHg and/or diastolic blood pressure ≥ 100 mmHg), with a history of hypertensive crisis or hypertensive encephalopathy.
12. Grade ≥ 2 peripheral neuropathy as per CTCAE 6.0.
13. Human immunodeficiency virus (HIV) infection.
14. Active pulmonary tuberculosis.
15. A history of or active interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonitis, or severe lung function impairment that may interfere with the detection and management of suspected drug-related pulmonary toxicity.
16. Known active or suspected autoimmune diseases. Patients with a history of autoimmune disease that does not require systemic immunosuppressive therapy for at least 12 months prior to screening are allowed to be enrolled.
17. Treatment with live vaccines within 28 days prior to randomization. Inactivated seasonal influenza vaccines and COVID-19 vaccines are allowed, but live attenuated influenza vaccines for intranasal use are not allowed.
18. Treatment with systemic glucocorticoids (> 10 mg/day prednisone efficacy dosage) or other immunosuppressive drugs required within 14 days prior to randomization or during the study. However, patients are allowed to be enrolled under the following conditions: in the absence of active autoimmune disease, patients are allowed to use topical or inhaled glucocorticoids and adrenal glucocorticoid replacement therapy at a dose equivalent to ≤ 10 mg/day of prednisone efficacy.
19. Any active infection requiring systemic anti-infective therapy or use of systemic anti-infective therapy within 14 days prior to randomization.
20. Major surgery within 28 days prior to randomization; major surgery in this study is defined as any surgery that requires at least 3 weeks of postoperative recovery time before receiving the study treatment. Patients with a history of tumor needle biopsy or lymph node incisional biopsy are allowed to be enrolled.
21. Radical radiotherapy within 3 months prior to randomization. Note: Palliative radiotherapy to bone or palliative radiotherapy to superficial lesions is allowed according to the local treatment guidelines, which should have been completed 2 weeks prior to randomization. Radiotherapy covering more than 30% of the bone marrow area within 28 days prior to randomization is not allowed.
22. Prior use of other antibodies/drugs against immune checkpoints, such as PD-1, PD-L1, CTLA4, etc. Patients with prior systemic anti-EGFR monoclonal antibody therapy.
23. Current participation in any other clinical study, or the end of the previous clinical study treatment is less than 14 days apart from the planned start of the study treatment in this study.
24. Known history of severe allergy to any monoclonal antibody.
25. Known allergy to any components of carboplatin or paclitaxel (or nab-paclitaxel).
26. Pregnant or lactating women.
27. Known history of psychotropic abuse or drug abuse; history of alcohol abuse.
28. Presence of any other factors that may lead to a premature study discontinuation as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2031-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
ORR assessed by BICR (part I) | Assessed up to appoximately 6 months from enrollment
  Defined as the proportion of participants who achieve a best overall response of CR or PR
PFS assessed by BICR (part I) | Assessed up to appoximately 16 months from enrollment
  Defined as the time from randomization to the first documentation of PD (RECIST v1.1) or death due to any cause (whichever occurs first)
PFS assessed by BICR (part II) | Assessed up to appoximately 23 months from enrollment
  Defined as the time from randomization to the first documentation of PD (RECIST v1.1) or death due to any cause (whichever occurs first)
OS (part II) | Assessed up to appoximately 42 months from enrollment
  Defined as the time from randomization to death due to any cause

SECONDARY OUTCOMES:
DCR (part I) | Assessed up to appoximately 6 months from enrollment
  Defined as the proportion of participants who achieve a best overall response of CR or PR or an SD
OS (part I) | Assessed up to appoximately 35 months from enrollment
  Defined as the time from randomization to death due to any cause
DOR (part I) | Assessed up to appoximately 35 months from enrollment
  Defined as the time from the first documented objective response to PD or death
ORR assessed by investigator (part I) | Assessed up to appoximately 6 months from enrollment
  Defined as the proportion of participants who achieve a best overall response of CR or PR
PFS assessed by investigator (part I) | Assessed up to appoximately 16 months from enrollment
  Defined as the time from randomization to the first documentation of PD (RECIST v1.1) or death due to any cause (whichever occurs first)
Incidence of adverse events (part I) | Assessed up to appoximately 35 months from enrollment
ORR (part II) | Assessed up to appoximately 6 months from enrollment
  Defined as the proportion of participants who achieve a best overall response of CR or PR
DCR (part II) | Assessed up to appoximately 6 months from enrollment
  defined as the proportion of participants who achieve a best overall response of CR or PR or an SD lasting for 12 weeks
DOR (part II) | Assessed up to appoximately 42 months from enrollment
  Defined as the time from the first documented objective response to PD or death
PFS assessed by investigator (part II) | Assessed up to appoximately 23 months from enrollment
  Defined as the time from randomization to the first documentation of PD (RECIST v1.1) or death due to any cause (whichever occurs first)
Incidence of adverse events (part II) | Assessed up to appoximately 42 months from enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No